CLINICAL TRIAL: NCT03233217
Title: Safety and Immunogenicity of High-Dose Quadrivalent Influenza Vaccine Administered by Intramuscular or Subcutaneous Route in Participants Aged 65 Years and Older in Japan
Brief Title: Safety and Immunogenicity of High-Dose Quadrivalent Influenza Vaccine in Patients ≥65 Years
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Collaborators: Sanofi (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: QHD00008; U1111-1183-5525 (Other: World Health Organization Universal Trial Number); DFI15130 (Other: Sanofi K.K.)
Record Dates: First submitted 2017-07-25; First posted 2017-07-28 (Actual); Results first posted 2019-12-17 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Influenza
Keywords: Influenza
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Intervention Model Description: Safety and tolerability was initially assessed in the first 10 participants in a smaller cohort (Cohort 1). Participants were randomized 1:1 into 2 groups in Cohort 1: QIV-HD by IM route (n=5) and QIV-HD by SC route (n=5).
  After review of the local and systemic adverse events, the remaining 165 participants were enrolled (Cohort 2). Participants were randomized 1:1:1 into 3 groups in Cohort 2: QIV-HD by IM route (n=55), QIV-HD by SC route (n=55), and QIV-SD by SC route (n=55).
Who Masked: Participant, Investigator
Masking Description: QHD00008 was a modified double-blind study in which only the designated administrator at each study site knew which vaccine was administered to the participants. The participants and the Investigator/Sub-investigator in charge of the safety assessment were blinded in order to decrease the potential bias in safety assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Cohort 1: QIV-HD by IM (Experimental): Participants were randomized to receive a single 0.7-milliliter (mL) injection of QIV-HD by IM route on Day 0.
  Interventions: Biological: QIV-HD by IM
- Cohort 1: QIV-HD by SC (Experimental): Participants were randomized to receive a single 0.7 mL injection of QIV-HD by SC route on Day 0.
  Interventions: Biological: QIV-HD by SC
- Cohort 2: QIV-HD by IM (Experimental): Participants were randomized to receive a single 0.7 mL injection of QIV-HD by IM route on Day 0.
  Interventions: Biological: QIV-HD by IM
- Cohort 2: QIV-HD by SC (Experimental): Participants were randomized to receive a single 0.7 mL injection of QIV-HD by SC route on Day 0.
  Interventions: Biological: QIV-HD by SC
- Cohort 2: QIV-SD by SC (Active Comparator): Participants were randomized to receive a single 0.5 mL injection of QIV-SD by SC route on Day 0.
  Interventions: Biological: QIV-SD by SC

INTERVENTIONS:
Biological: QIV-HD by IM — IM, injected into the upper arm (deltoid area)
  Other Names: High-Dose Influenza Vaccine Quadrivalent (IM)
  Arms: Cohort 1: QIV-HD by IM; Cohort 2: QIV-HD by IM
Biological: QIV-SD by SC — SC, injected into the upper arm (posterior region)
  Other Names: Standard-Dose Influenza Vaccine Quadrivalent
  Arms: Cohort 2: QIV-SD by SC
Biological: QIV-HD by SC — SC, injection into the upper arm (posterior region)
  Other Names: High-Dose Influenza Vaccine Quadrivalent (SC)
  Arms: Cohort 1: QIV-HD by SC; Cohort 2: QIV-HD by SC

SUMMARY:
This phase I/II, randomized, modified double-blind, multi-center study assessed the safety and immunogenicity of a high-dose Quadrivalent influenza vaccine (QIV-HD) in older adults (greater than or equal to [>=] 65 years).

DETAILED DESCRIPTION:
This phase I/II, randomized, modified double-blind, multi-center study was conducted in 175 healthy Japanese adults aged 65 years and older to describe the safety profile and immune responses (geometric mean titers and seroconversion for the 4 common strains at 28 days post-vaccination) of the QIV-HD administered by intramuscular (IM) and subcutaneous (SC) methods. A local standard-dose Quadrivalent Influenza Vaccine (QIV-SD) administered by SC method served as a control arm.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 65 years on the day of inclusion.
* Informed consent form has been signed and dated.
* Able to attend all scheduled visits and to comply with all study procedures.

Exclusion Criteria:

* Participation at the time of study enrollment (or in the 4 weeks preceding the study vaccination) or planned participation during the present study period in another clinical study investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccination with live vaccines within the past 27 days preceding the study vaccination or any vaccination with inactivated vaccines within the past 6 days preceding the study vaccination, or planned receipt of any vaccine prior to Visit 3.
* Previous vaccination against influenza (in the preceding 6 months) with either the study vaccine or another vaccine.
* Receipt of immune globulins, blood or blood-derived products in the past 3 months.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy, within the preceding 6 months; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks within the past 3 months).
* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components, or history of a life-threatening reaction to the vaccine used in the study or to a vaccine containing any of the same substances.
* Thrombocytopenia or bleeding disorder, contraindicating IM vaccination based on Investigator's judgment.
* Deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized involuntarily.
* Alcohol or substance abuse that, in the opinion of the Investigator might interfere with the study conduct or completion.
* Chronic illness that, in the opinion of the Investigator, was at a stage where it might interfere with study conduct or completion.
* Identified as an Investigator or employee of the Investigator or study center with direct involvement in the proposed study, or identified as an immediate family member (i.e., parent, spouse, natural or adopted child) of the Investigator or employee with direct involvement in the proposed study.
* Personal or family history of Guillain-Barré syndrome.
* Neoplastic disease or any hematologic malignancy (except localized skin or prostate cancer that was stable at the time of vaccination in the absence of therapy and participants who had a history of neoplastic disease and have been disease free for >=5 years).
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >=37.5°Celsius). A prospective participant were not be included in the study until the condition had resolved or the febrile event had subsided.
* History of convulsions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 175 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (2):
- Japan (2):
  - Sanofi Pasteur Investigational Site, Ōsaka
  - Sanofi Pasteur Investigational Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

REFERENCES:
- [Background] Sanchez L, Matsuoka O, Inoue S, Inoue T, Meng Y, Nakama T, Kato K, Pandey A, Chang LJ. Immunogenicity and safety of high-dose quadrivalent influenza vaccine in Japanese adults >/=65 years of age: a randomized controlled clinical trial. Hum Vaccin Immunother. 2020 Apr 2;16(4):858-866. doi: 10.1080/21645515.2019.1677437. Epub 2019 Nov 19. PMID 31634025
- See also: Related info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 15 September 2017 to 26 October 2017 at 2 centers in Japan.
Pre-assignment Details: 10 participants were randomized 1:1 to receive either QIV-HD by intramuscular (IM) route or QIV-HD by subcutaneous (SC) route (Cohort 1). After review of local and systemic AEs for 7 days post-vaccination in Cohort 1, remaining 165 participants were randomized 1:1:1 to receive QIV-HD by IM route, QIV-HD by SC route, or QIV-SD by SC route (Cohort 2)
Groups:
- Cohort 1: QIV-HD by IM: Participants were randomized to receive a single 0.7-milliliter (mL) injection of high-dose Quadrivalent influenza vaccine (QIV-HD) by IM route on Day 0.
- Cohort 2: QIV-SD by SC: Participants were randomized to receive a single 0.5 mL injection of standard-dose Quadrivalent influenza vaccine (QIV-SD) by SC route on Day 0.
Period: Overall Study
Arm/Group | Cohort 1: QIV-HD by IM | Cohort 1: QIV-HD by SC | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Started (Randomized and vaccinated.) | 5 | 5 | 55 | 55 | 55
Safety Analysis Set (SafAS) | 5 | 5 | 55 | 55 | 55
Per-protocol Analysis Set (PPAS) (Cohort 1 = 10 participants, and Cohort 2 = 164 participants) | 5 | 5 | 55 | 55 | 54
Completed | 5 | 5 | 55 | 55 | 55
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The baseline characteristics was analyzed on SafAS which included participants who received study vaccine and analyzed according to the vaccine they actually received.
Groups:
- Cohort 1: QIV-HD by IM; Cohort 2: QIV-HD by IM: Participants were randomized to receive a single 0.7 mL injection of QIV-HD by IM route on Day 0.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: QIV-HD by IM | Cohort 1: QIV-HD by SC | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC | Total
Number analyzed (Participants) | 5 | 5 | 55 | 55 | 55 | 175
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.8 (2.0) | 70.8 (2.3) | 70.1 (3.7) | 70.5 (3.6) | 69.9 (3.8) | 70.2 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 27 | 26 | 25 | 80
  Male | 4 | 4 | 28 | 29 | 30 | 95
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 5 | 55 | 55 | 55 | 175
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Unsolicited Adverse Events (AE) After Vaccination
Description: An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of symptom and/or onset post-vaccination. Unsolicited AEs includes both serious and non-serious unsolicited AEs. A serious adverse event is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event. All participants were observed for 30 minutes after vaccination, and any unsolicited AEs occurred during that time were recorded as immediate unsolicited AEs in the CRB.
Time Frame: Within 30 minutes after vaccination
Population: The safety analysis was performed on SafAS which included participants who received study vaccine and analyzed according to the vaccine they actually received. Data for this outcome measure was planned to be collected and analyzed for combined population of Cohort 1 and Cohort 2 participants who received QIV-HD (QIV-HD by IM and QIV-HD by SC).
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1 and 2: QIV-HD by IM: Participants were randomized to receive a single 0.7 mL injection of QIV-HD by IM route on Day 0.
- Cohort 1 and 2: QIV-HD by SC: Participants were randomized to receive a single 0.7 mL injection of QIV-HD by SC route on Day 0.
Arm/Group | Cohort 1 and 2: QIV-HD by IM | Cohort 1 and 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 60 | 60 | 55
Participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Solicited Injection Site and Systemic Reactions
Description: A solicited reaction was an adverse reaction observed and reported under the conditions (symptom and onset) prelisted (i.e., solicited) in the CRB and considered as related to the administered vaccination. Solicited injection site reactions: pain, erythema, swelling, induration, and bruising. Solicited systemic reactions: fever, headache, malaise, myalgia, and shivering.
Time Frame: Within 7 days after vaccination
Population: The safety analysis was performed on SafAS which included participants who received study vaccine and analyzed according to the vaccine they actually received. Data for this outcome measure was planned to be collected and analyzed for combined population for Cohort 1 and Cohort 2 participants who received QIV-HD (QIV-HD by IM and QIV-HD by SC).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: QIV-HD by IM | Cohort 1 and 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 60 | 60 | 55
Participants
  Injection site pain | 18 | 27 | 15
  Injection site erythema | 11 | 19 | 11
  Injection site swelling | 9 | 17 | 13
  Injection site induration | 2 | 7 | 2
  Injection site bruising | 0 | 0 | 0
  Fever | 0 | 1 | 0
  Headache | 3 | 8 | 1
  Malaise | 1 | 4 | 3
  Myalgia | 9 | 16 | 7
  Shivering | 0 | 2 | 2

3. Primary Outcome: Number of Participants With Unsolicited Adverse Events After Vaccination
Description: An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the CRB in terms of symptom and/or onset post-vaccination. Unsolicited AEs included both serious and non-serious unsolicited AEs. A serious adverse event is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Within 28 days after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: QIV-HD by IM | Cohort 1 and 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 60 | 60 | 55
Participants | 4 | 4 | 8

4. Primary Outcome: Number of Participant With Serious Adverse Events (SAEs) After Vaccination
Description: An SAE is any untoward medical occurrence that at any dose results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, or is an important medical event.
Time Frame: Up to 6 months after vaccination
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 and 2: QIV-HD by IM | Cohort 1 and 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 60 | 60 | 55
Participants | 0 | 0 | 1

5. Secondary Outcome: Cohort 2: Geometric Mean Titers (GMTs) of Influenza Antibodies Following Vaccination With QIV-HD or QIV-SD
Description: GMT of anti-influenza antibodies strains (A1, A1-like, A2, A2-like, B1, B2, B2-like) were measured using a hemagglutination inhibition (HAI) assay.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: Analyzed on PPAS which included all participants who received at least 1 dose of study vaccine, and had post-vaccination blood sample HAI result for at least 1 strain, with no protocol deviations. Here, 'number analyzed' = participants with available data for each category. Data for this outcome measure was not planned to be analyzed for Cohort 1.
Measure: Geometric Mean (95% Confidence Interval); unit: titers (1/dilution)
Arm/Group | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 55 | 55 | 54
titers (1/dilution)
  A1: Day 0 | 44.5 [29.4 to 67.5] | 59.5 [39.7 to 89.2] | 41.0 [27.7 to 60.8]
  A1-like: Day 0: number analyzed (Participants) | 55 | 55 | 53
  A1-like: Day 0 | 46.2 [35.4 to 60.4] | 56.2 [43.0 to 73.5] | 42.1 [32.8 to 54.1]
  A2: Day 0 | 62.6 [39.9 to 98.1] | 101.0 [66.9 to 152.6] | 83.7 [53.9 to 129.9]
  A2-like: Day 0 | 76.1 [49.6 to 116.7] | 107.6 [71.4 to 162.1] | 91.0 [57.7 to 143.3]
  B1: Day 0 | 116.8 [83.2 to 163.9] | 134.1 [92.2 to 195.0] | 108.2 [79.5 to 147.1]
  B2: Day 0 | 76.1 [49.9 to 115.9] | 109.6 [73.4 to 163.8] | 97.6 [69.6 to 137.0]
  B2-like: Day 0 | 32.7 [22.9 to 46.7] | 47.1 [32.8 to 67.6] | 41.6 [31.4 to 55.1]
  A1: Day 28 | 712.4 [509.7 to 995.7] | 550.2 [402.2 to 752.5] | 269.1 [181.5 to 399.0]
  A1-like: Day 28 | 427.6 [309.1 to 591.5] | 356.2 [260.0 to 488.0] | 216.3 [157.4 to 297.3]
  A2: Day 28 | 1059.5 [759.5 to 1478.0] | 839.2 [617.7 to 1140.0] | 405.8 [270.5 to 608.6]
  A2-like: Day 28: number analyzed (Participants) | 55 | 55 | 53
  A2-like: Day 28 | 940.0 [664.3 to 1330.1] | 797.9 [586.8 to 1084.9] | 402.3 [263.0 to 615.4]
  B1: Day 28 | 877.0 [632.9 to 1215.3] | 628.0 [475.4 to 829.6] | 336.9 [263.7 to 430.3]
  B2: Day 28 | 813.2 [603.0 to 1096.5] | 758.7 [589.5 to 976.5] | 281.5 [217.0 to 365.0]
  B2-like: Day 28 | 269.9 [199.4 to 365.4] | 261.6 [201.1 to 340.2] | 111.0 [87.6 to 140.7]

6. Secondary Outcome: Cohort 2: Geometric Mean Titer Ratios (GMTRs) of Influenza Antibodies Following Vaccination With QIV-HD or QIV-SD
Description: GMT of anti-influenza antibodies strains (A1, A1-like, A2, A2-like, B1, B2, B2-like) were measured using an HAI assay. GMTRs were calculated as the ratio of GMTs post vaccination and pre-vaccination.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: The analysis was performed on PPAS which included all participants who received at least 1 dose of study vaccine, and had post-vaccination blood sample HAI result for at least 1 strain, with no protocol deviations. Data for this outcome measure was not planned to be analyzed for Cohort 1.
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 55 | 55 | 54
ratio
  A1: Day 28/Day 0 | 16.00 [10.19 to 25.11] | 9.25 [6.11 to 14.00] | 6.56 [4.36 to 9.86]
  A1-like: Day 28/Day 0 | 9.25 [6.67 to 12.82] | 6.34 [4.79 to 8.38] | 5.13 [3.67 to 7.17]
  A2: Day 28/Day 0 | 16.93 [10.99 to 26.10] | 8.31 [5.54 to 12.46] | 4.85 [3.08 to 7.63]
  A2-like: Day 28/Day 0 | 12.36 [8.03 to 19.01] | 7.42 [4.98 to 11.05] | 4.56 [2.89 to 7.19]
  B1: Day 28/Day 0 | 7.51 [4.93 to 11.45] | 4.68 [3.34 to 6.56] | 3.11 [2.29 to 4.24]
  B2: Day 28/Day 0 | 10.69 [7.05 to 16.21] | 6.92 [4.79 to 9.99] | 2.88 [2.08 to 3.99]
  B2-like: Day 28/Day 0 | 8.26 [5.74 to 11.89] | 5.55 [3.97 to 7.76] | 2.67 [2.00 to 3.57]

7. Secondary Outcome: Cohort 2: Percentage of Participants Achieving Seroconversion Against Antigens Following Vaccination With QIV-HD or QIV-SD
Description: Anti-influenza antibodies were measured by using the HAI assay for the strains A1, A1-like, A2, A2-like, B1, B2, and B2-like. Seroconversion was defined as either a HAI titer lesser than (<) 10 (1/dilution) at Day 0 and post-vaccination titer greater than or equal to (>=) 40 (1/dilution) at Day 28, or HAI titer >=10 (1/dilution) at Day 0 and a >=4-fold increase in HAI titer (1/dilution) at Day 28.
Time Frame: Day 28 (post-vaccination)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 55 | 55 | 54
percentage of participants
  A1 | 74.5 [61.0 to 85.3] | 67.3 [53.3 to 79.3] | 55.6 [41.4 to 69.1]
  A1-like: number analyzed (Participants) | 55 | 55 | 53
  A1-like | 74.5 [61.0 to 85.3] | 69.1 [55.2 to 80.9] | 56.6 [42.3 to 70.2]
  A2 | 85.5 [73.3 to 93.5] | 63.6 [49.6 to 76.2] | 42.6 [29.2 to 56.8]
  A2-like: number analyzed (Participants) | 55 | 55 | 53
  A2-like | 74.5 [61.0 to 85.3] | 58.2 [44.1 to 71.3] | 43.4 [29.8 to 57.7]
  B1 | 58.2 [44.1 to 71.3] | 47.3 [33.7 to 61.2] | 37.0 [24.3 to 51.3]
  B2 | 65.5 [51.4 to 77.8] | 63.6 [49.6 to 76.2] | 33.3 [21.1 to 47.5]
  B2-like | 67.3 [53.3 to 79.3] | 60.0 [45.9 to 73.0] | 33.3 [21.1 to 47.5]

8. Secondary Outcome: Cohort 2: Percentage of Participants Achieving Seroprotection Against Antigens Following Vaccination With QIV-HD or QIV-SD
Description: Anti-influenza antibodies were measured by using the HAI assay for the strains A1, A1-like, A2, A2-like, B1, B2, and B2-like. Seroprotection was defined as a HAI titer >=40 (1/dilution) at Day 0 and Day 28.
Time Frame: Day 0 (pre-vaccination) and Day 28 (post-vaccination)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 2: QIV-HD by IM | Cohort 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
Number analyzed (Participants) | 55 | 55 | 54
percentage of participants
  A1: Day 0 | 60.0 [45.9 to 73.0] | 65.5 [51.4 to 77.8] | 53.7 [39.6 to 67.4]
  A1-like: Day 0: number analyzed (Participants) | 55 | 55 | 53
  A1-like: Day 0 | 58.2 [44.1 to 71.3] | 60.0 [45.9 to 73.0] | 54.7 [40.4 to 68.4]
  A2: Day 0 | 63.6 [49.6 to 76.2] | 83.6 [71.2 to 92.2] | 68.5 [54.4 to 80.5]
  A2-like: Day 0 | 65.5 [51.4 to 77.8] | 81.8 [69.1 to 90.9] | 70.4 [56.4 to 82.0]
  B1: Day 0 | 76.4 [63.0 to 86.8] | 87.3 [75.5 to 94.7] | 81.5 [68.6 to 90.7]
  B2: Day 0 | 67.3 [53.3 to 79.3] | 78.2 [65.0 to 88.2] | 79.6 [66.5 to 89.4]
  B2-like: Day 0 | 49.1 [35.4 to 62.9] | 52.7 [38.8 to 66.3] | 57.4 [43.2 to 70.8]
  A1: Day 28 | 98.2 [90.3 to 100.0] | 100 [93.5 to 100.0] | 92.6 [82.1 to 97.9]
  A1-like: Day 28 | 98.2 [90.3 to 100.0] | 100 [93.5 to 100.0] | 98.1 [90.1 to 100.0]
  A2: Day 28 | 100 [93.5 to 100.0] | 100 [93.5 to 100.0] | 96.3 [87.3 to 99.5]
  A2-like: day 28: number analyzed (Participants) | 55 | 55 | 53
  A2-like: day 28 | 100 [93.5 to 100.0] | 100 [93.5 to 100.0] | 96.2 [87.0 to 99.5]
  B1: Day 28 | 98.2 [90.3 to 100.0] | 100 [93.5 to 100.0] | 98.1 [90.1 to 100.0]
  B2: Day 28 | 98.2 [90.3 to 100.0] | 100 [93.5 to 100.0] | 98.1 [90.1 to 100.0]
  B2-like: Day 28 | 98.2 [90.3 to 100.0] | 100 [93.5 to 100.0] | 94.4 [84.6 to 98.8]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data was collected from Day 0 (post-vaccination) up to Day 28 after vaccination. Solicited Reaction (SR) data were collected up to Day 7 after vaccination. Serious adverse event (SAE) data were collected throughout the study (up to 28 days after vaccination).
Description: Analyzed on SafAS. SR: an AE prelisted in CRB and considered related to vaccination. SR was therefore an adverse reaction observed and reported under conditions (symptom and onset) prelisted in CRB. An unsolicited AE: an observed AE that did not fulfill conditions prelisted in CRB in terms of symptom and/or onset post-vaccination. AE data were planned to be collected and analyzed for the combined population of Cohort 1 and Cohort 2 participants who received QIV-HD (QIV-HD by IM and QIV-HD by SC)
Arm/Group | Cohort 1 and 2: QIV-HD by IM | Cohort 1 and 2: QIV-HD by SC | Cohort 2: QIV-SD by SC
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 1/55
Other Adverse Events (participants affected / at risk) | 4/60 | 4/60 | 7/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: QIV-HD by IM (N=60) | Cohort 1 and 2: QIV-HD by SC (N=60) | Cohort 2: QIV-SD by SC (N=55)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 and 2: QIV-HD by IM (N=60) | Cohort 1 and 2: QIV-HD by SC (N=60) | Cohort 2: QIV-SD by SC (N=55)
Cystitis (Infections and infestations) | 1 | 0 | 0
Laryngitis (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 2 | 2
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Faeces soft (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Injection site pruritus (General disorders) | 1 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2017-05-12): https://cdn.clinicaltrials.gov/large-docs/17/NCT03233217/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-13): https://cdn.clinicaltrials.gov/large-docs/17/NCT03233217/SAP_001.pdf